CLINICAL TRIAL: NCT03064750
Title: Pelvic Floor Exercise Before Surgery in Women With Pelvic Organ Prolapse
Acronym: CONTRAPOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1751
Record Dates: First submitted 2017-02-22; First posted 2017-02-27 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Pelvic Organ Prolapse; Pelvic Floor Disorders
Keywords: Exercise Therapy; Pelvic Floor; Preoperative Care
MeSH Terms: conditions — Pelvic Organ Prolapse; Pelvic Floor Disorders | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-surgery exercise (Experimental): pelvic floor exercises individually and in groups
  Interventions: Behavioral: pelvic floor exercises
- Waiting list (Other): wait as usual until surgery
  Interventions: Other: Waiting list

INTERVENTIONS:
Behavioral: pelvic floor exercises — In preparation for surgery, patients receive individual information by a physiotherapist on pelvic floor anatomy and correct pelvic floor contraction. Patients are told to do the following pelvic floor exercises 3 times a day: 8-12 maximal contractions, hold contractions during 10 seconds, and 3 fast contractions after each long contraction. In addition exercise in groups with skilled physical therapists once a week during 12 weeks.
  Arms: Pre-surgery exercise
Other: Waiting list — patients wait as usual until surgery without special treatment.
  Arms: Waiting list

SUMMARY:
The lifetime risk for a woman to undergo surgery for either vaginal prolapse or urinary incontinence is high. There are many different surgical techniques for treatment of prolapse, but there is a lack of knowledge about factors that contribute to objective result and patient satisfaction after surgery.

The aim of the study is to investigate factors that could be related to patient satisfaction and objective result such as pelvic floor muscle contractility/strength and muscle injury, objective measures of prolapse and women's symptoms. This study will investigate whether systematic pelvic floor exercise and life style advise before surgery can improve outcomes after surgery for either vaginal prolapse. Another aim is to determine an ultrasound scale for measure of pelvic floor muscle contraction.

ELIGIBILITY:
Inclusion Criteria:

* referred to surgery for urogenital prolapse
* informed consent

Exclusion Criteria:

* not able to communicate in Norwegian or English
* not able or willing to sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle strength assessed by palpation | 9 months
  Muscle strength is evaluated using 6 point modified Oxford Scale (MOS) range 0-5.
Pelvic floor muscle strength assessed by ultrasound | 9 months
  Changes in pelvic floor muscle at rest and during pelvic floor contraction, measured in mm and calculated proportional change
Symptoms of pelvic floor disorders | 9 months
  Symptoms of pelvic floor disorders assessed by validated questionnaire (PDFI-20)

SECONDARY OUTCOMES:
Pelvic floor muscle strength assessed by perineometry | 9 months
  measuring the pressure with vaginal manometry in cm H2O during pelvic floor contraction
Pelvic floor muscle strength assessed by electromyography | 9 months
  Assessed by vaginal surface electrode during pelvic floor contraction, measured in mV
Proportion of anatomical pelvic organ prolapse | 9 months
  Assessment with the Pelvic Organ Prolapse Quantification (POP-Q) System
Proportion of anatomical sphincter ani defect | 9 months
  Anatomical sphincter ani defect assessed by transperineal ultrasound
Proportion of levator ani muscle trauma | 9 months
  Assessed by transperineal ultrasound on contraction and Valsalva
Assessment of pelvic organ mobility as a measure of pelvic organ function/dysfunction | 9 months
  Movement of the pelvic organs during Valsalva and contraction
Imaging of synthetic implants assessed by ultrasound | 9 months
  Registration of implants after pelvic floor surgery and their relations to anatomical structures in mm.
Symptoms of pelvic floor disorders | 9 months
  Symptoms of pelvic floor disorders assessed by validated questionnaire (PFIQ-7)
Symptoms of pelvic floor disorders | 9 months
  Symptoms of pelvic floor disorders assessed by visual analogue scale (VAS 1-10)

CONTACTS AND LOCATIONS:
Overall Officials: Kjell Å Salvesen, md prof, Study Director — St Olavs Hospital University Hospital Trondheim
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nyhus MO, Oversand SH, Salvesen O, Salvesen KA, Mathew S, Volloyhaug I. Ultrasound assessment of pelvic floor muscle contraction: reliability and development of an ultrasound-based contraction scale. Ultrasound Obstet Gynecol. 2020 Jan;55(1):125-131. doi: 10.1002/uog.20382. Epub 2019 Dec 13. PMID 31237722
- [Result] Nyhus MO, Mathew S, Salvesen O, Salvesen KA, Stafne S, Volloyhaug I. Effect of preoperative pelvic floor muscle training on pelvic floor muscle contraction and symptomatic and anatomical pelvic organ prolapse after surgery: randomized controlled trial. Ultrasound Obstet Gynecol. 2020 Jul;56(1):28-36. doi: 10.1002/uog.22007. Epub 2020 Jun 9. PMID 32144829
- [Result] Mathew S, Nyhus MO, Salvesen O, Salvesen KA, Stafne SN, Volloyhaug I. The effect of preoperative pelvic floor muscle training on urinary and colorectal-anal distress in women undergoing pelvic organ prolapse surgery-a randomized controlled trial. Int Urogynecol J. 2021 Oct;32(10):2787-2794. doi: 10.1007/s00192-021-04684-3. Epub 2021 Feb 13. PMID 33580809